CLINICAL TRIAL: NCT03398772
Title: Effects of a Comprehensive Health Coaching Program on Lung Function, Exercise Tolerance, Symptom Distress, Quality of Life, Readmission, and Survival in Advanced Chronic Obstructive Pulmonary Disease Patients: A Randomized Controlled Trial.
Brief Title: Effects of a Comprehensive Health Coaching Program in Advanced Chronic Obstructive Pulmonary Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201704032
Record Dates: First submitted 2018-01-02; First posted 2018-01-12 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2017-11

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe; Chronic Obstructive Pulmonary Disease End Stage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Comprehensive Health Coaching Program
  Interventions: Behavioral: Comprehensive Health Coaching Program
- Control (No Intervention): Guideline-based usual care

INTERVENTIONS:
Behavioral: Comprehensive Health Coaching Program — Comprehensive Health Coaching Program: included physical activity and motivational interviewing techniques, participants were encouraged to set goals with decision-making, self-management and self-monitor their progress, and received support from researcher.
  Arms: Experiment

SUMMARY:
Chronic obstructive pulmonary disease due to incurable and prevalence has increased steadily, chronic respiratory disease is considered hazardous to health and quality of life of the disease. GOLD treatment guidelines (global initiative for chronic obstructive lung disease guideline) pointed out the pulmonary rehabilitation is one of the non-drug treatment in patients with severe COPD, shown to improve exercise capacity and reduce the short of breathing, improve the quality of life and reduce the anxiety associated and depression and improved survival advantages. Meanwhile, a few studies have examined effect the exercise training in severe COPD patients' symptom distress and quality of life, so as to make severe COPD patients to improve the effectiveness of the campaign to ongoing regular pulmonary rehabilitation movement, is considered an important issue.

It has been proposed that physical activity enhancement or exercise training can be effective in improving symptoms and quality of life in these patients. However, it has not been examined systematically. Therefore, the main purposes of this study are: 1.Prevalence of symptom distress; 2.The physical preferences; 3.The relationship between quality of life and physical activity; 4.Effects of Comprehensive Health coaching exercise training on improving fatigue, sleep disturbances, quality of life, readmission, and survival. In the first year of this study, a descriptive-correlational design will be used and in the second and third years of study, the experimental design and prospective longitudinal study will be undertaken. Instruments include motion sensors, physical activity scale, Physical Activity Preferences, Pittsburgh Sleep Quality of Life Index. Statistical analyses include descriptive statistics, t-test, one-way ANOVA, latent growth modeling, Logistic models, GEE, and survival analysis. Results from this study will provide important implications for improving symptom management and quality of life for sever chronic obstructive pulmonary disease patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥40 years and ≦80 years
* patients with advanced COPD are defined according to the diagnostic criteria for severe (GOLD 3) and very severe (GOLD 4)
* pulmonologist assess need pulmonary rehabilitation, but not accept any rehabilitation exercise program.
* pulmonologist assessment the patients with a stable state.
* awareness, has the ability to read, write, and communication.
* willing to communicate by phone, and can operate smart phones.

Exclusion Criteria:

* COPD AE requiring corticosteroids, antibiotics, emergency room visit or hospitalization within the past 3 month.
* diagnosed mentally or cognitive disorder, such as dementia or unable to cooperate.
* severe hip, knee disease, can not perform exercise, or with neuromuscular dysfunction, such as limb hemiplegia, no independent walking function or other deterioration due to bone and joint disease.
* combined with severe heart disease, such as AMI, severe arrhythmia or heart failure.
* current regular practice of physical activity

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Lung function at 3 months, 6months | 3 months, 6months
  Spirometry (FEVl % predicted )
Change from Baseline Exercise Tolerance at 3 months, 6months | 3 months, 6months
  6 Minute walking test

SECONDARY OUTCOMES:
Change from Baseline Health-related quality of life at 3 months, 6months | 3 months, 6months
  St. George's Respiratory Questionnaire
Change from Baseline Fatigue at 3 months, 6months | 3 months, 6months
  Brief Fatigue Inventory Short Form BFI-Taiwan Form
Change from Baseline Psychological distress at 3 months, 6months | 3 months, 6months
  Hospital Anxiety and Depression Scale
Change from Baseline Symptom Distress at 3 months, 6months | 3 months, 6months
  Taiwanese version of the M. D. Anderson Symptom Inventory
Change from Baseline Quality of Sleep at 3 months, 6months | 3 months, 6months
  Taiwanese version of the Pittsburgh Sleep Quality Index
Readmission rate Survival | 1 year
  pulmonologists blinded to allocation reviewed admission summaries and information to determine as COPD related readmission or mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical Hospital-Shuang Ho Hospital,Ministry of Health and Welfare, Taipei, Taiwan